CLINICAL TRIAL: NCT01739426
Title: Evaluation of Endoscopic Treatment of Zenker's Diverticulum Using the LigaSure Thermal Vessel Sealing System
Brief Title: Evaluation of Endoscopic Treatment of Zenker's Diverticulum Using LigaSure
Acronym: ZENKER LS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2012/SK-02; 2012-A01096-37 (Other: RCB number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-03 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Zenker Diverticulum
Keywords: LigaSure V (TM)
MeSH Terms: conditions — Zenker Diverticulum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study population (Experimental): The population is composed of patients with a confirmed Zenker's diverticulum.
  Intervention: Repair w/LigaSure
  Interventions: Device: Repair w/LigaSure

INTERVENTIONS:
Device: Repair w/LigaSure — Surgical repair is carried out as normal except that a novel device is used: LigaSure V (TM) laparoscopic instrument (reference LS1500)

SUMMARY:
The primary objective of this study is to evaluation the success of endoscopic treatment of Zenker's diverticulum using a LigaSure device (thermal fusion of vessels) via a measure of swallowing function at 12 months post-surgery.

DETAILED DESCRIPTION:
Our secondary objectives are:

A. To evaluate short-term (pain, fever, time to start of eating) and medium-term (weight, swallowing) post-operative parameters.

B. To evaluate the prevalence of post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* The patient has a Zenkers diverticulum as confirmed by a pharyngo-oesophagean transit test, regardless of van Overbeek classification

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient (or his/her person-of-trust) refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient does not read french
* The patient is pregnant
* The patient is breastfeeding
* The patients has a contraindication for a treatment necessary for this study, or for general anesthesia
* The patent has a history of complications related to hemostasis
* The preoperative checkup indicates potential for hemostasis related problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Operational success according to the van Overbeek classification (yes/no) | 12 months
Change in Deglutition Handicap Index score | baseline to 12 months

SECONDARY OUTCOMES:
Change in Deglutition Handicap Index score | baseline to Day 3
Change in Deglutition Handicap Index score | baseline to 6-8 weeks
Change in visual analog scale for pain | baseline to day 1
  Visual analog scale varying from 0 to 10
Change in visual analog scale for pain | baseline to day 2
  Visual analog scale varying from 0 to 10
Change in visual analog scale for pain | baseline to day 3
  Visual analog scale varying from 0 to 10
Change in Temperature (°C) | baseling to Day 1
Change in Temperature (°C) | baseling to Day 2
Change in Temperature (°C) | baseling to Day 3
Time until the patient restarts eating (hours) | Day 1
Time until the patient restarts eating (hours) | Day 2
Time until the patient restarts eating (hours) | Day 3
Change in weight | baseline to 6-8 weeks
  Change in weight measured in kilograms
Change in weight | baseline to 12 months
  Change in weight measured in kilograms
Presence/absence of post-operative complications | Day 0 (day of surgery)
Presence/absence of post-operative complications | Day 1
Presence/absence of post-operative complications | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Kacha, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France